CLINICAL TRIAL: NCT03090698
Title: Viscosupplementation in Patients With Severe Osteoarthritis of the Knee
Brief Title: Outcomes of Injections in Patients Waiting for Total Knee Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Vinicius Schott Gameiro, Clinical Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VISCO KNEE UFF
Record Dates: First submitted 2017-03-02; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; treatment
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — hylan; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Hylan (Active Comparator): Intra-articular (knee) 6ml Hylan GF20 administration (single shot)
  Interventions: Drug: Hylan G-F 20
- Hylan + Corticosteroid (Active Comparator): Intra-articular (knee) 6ml Hylan GF20 and 1ml Triamcinolone 20mg/ml administration (single shot)
  Interventions: Drug: Hylan G-F 20; Drug: Triamcinolone
- Corticosteroid (Active Comparator): Intra-articular (knee) 1ml Triamcinolone administration (single shot)
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Hylan G-F 20 — intra-articular administration
  Arms: Hylan; Hylan + Corticosteroid
Drug: Triamcinolone — Intra-articular administration
  Arms: Corticosteroid; Hylan + Corticosteroid

SUMMARY:
A comparison of intraarticular administration of Hylan GF20, Triamcinolone and both associated in patients with severe osteoarthritis of the knee with follow up of one, three and six months.

DETAILED DESCRIPTION:
The objective of this research is to evaluate the short-term results of viscosupplementation in patients with advanced osteoarthritis of the knee.

There is a bigger demand of patients requiring total knee arthroplasty than the number of surgeries performed by the Unified Health System in Brazil. For this reason the queues to perform this surgery are huge and time-consuming in the referral hospitals. Whereas all these patients are suffering from severe pain and limiting, and awaiting the surgery for a few years, it is necessary to try any treatment, even if temporary, to ease the pain and suffering of those patients.

A double-blind randomized prospective study will be held at Hospital Federal dos Servidores do Estado do Rio de Janeiro, with patients from the waiting list for Total Knee Arthroplasty who accept to participate and sign the informed consent form. Will be selected the last 150 knees in TKA queue. Patients will be randomized and divided in 3 groups of 50 knees. A group will be submitted to an intraarticular injection of corticosteroid (1 ml of sterile Triamcinolone Hexacetonide solution 20 mg/ml). A second group will be subjected to administration of 6 ml of Hylan GF20. The third group will receive Hylan GF20 associated with corticosteroid (7 ml solution containing 1 ml of triamcinolone and 6 ml of Hylan GF20). The injection technique will be the same for all patients. The outcome results will be measured by a form with patient data, functional scores (Knee Society Score and Lysholm) before treatment and at one, three and six months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Waiting for Total Knee Arthroplasty (at Hospital Federal dos Servidores queue);
* Acceptance and signature of the TFCC;

Exclusion Criteria:

* Infiltration of the knee for the past 6 months;
* Allergic to any substance used in the study;
* Prior infection in the knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Lysholm M1 | One month
  The outcome will be measured by Lysholm Score within one month. The results will be compared within each group from baseline and between the 3 groups.
KSS M1 | One month
  The outcome will be measured by Knee Society Score within one month. The results will be compared within each group from baseline and between the 3 groups.

SECONDARY OUTCOMES:
Lysholm M3 | Three months
  The outcome will be measured by Lysholm Score within three months. The results will be compared within each group from baseline and between the 3 groups.
KSS M3 | Three months
  The outcome will be measured by Knee Society Score within three months. The results will be compared within each group from baseline and between the 3 groups.
Lysholm M6 | Six months
  The outcome will be measured by Lysholm Score within six months. The results will be compared within each group from baseline and between the 3 groups.
KSS M6 | Six months
  The outcome will be measured by Knee Society Score within six months. The results will be compared within each group from baseline and between the 3 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Campos, Principal Investigator — Hospital dos Servidores do Estado
Locations (1):
- Hospital dos Servidores do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided